CLINICAL TRIAL: NCT05740410
Title: Retrospective Analysis for the ClotTriever Catheter to Investigate Safety and Effectiveness in the Treatment of Acute and Subacute Iliofemoral Deep Vein Thrombosis (DVT)
Status: Completed | Type: Observational
Sponsor: Klinikum Arnsberg (Other)
Responsible Party: Sponsor
Other Study IDs: ClotTriever
Record Dates: First submitted 2023-01-30; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ClotTriever Catheter — Treatment of iliofemoral deep vein thrombosis with the ClotTriever catheter

SUMMARY:
The aim of the study is to evaluate the safety and performance of the ClotTriever catheter in the treatment of patients with symptomatic iliofemoral deep vein thrombosis (DVT)

DETAILED DESCRIPTION:
Data from patients in whom the ClotTriever catheter was used for treatment of iliofemoral DVT was retrospectively collected for up to 6 months after the procedure for evaluation of safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* uni or bilateral iliofemoral DVT

Exclusion Criteria:

* previously stented in treatment vein

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients treated in the vascular center of the clinic
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Procedural success | directly after treatment of the vein (Day 0)
  Restauration of inflow in the treated vein

SECONDARY OUTCOMES:
Incidence of ClotTriever related major adverse events (MAE) | 1 month
  MAEs defined as death, major amputation or any clinically driven target lesion revascularisation
Number of lesions with at least Society Interventional Radiology (SIR) Grad II Lyse (50-95% thrombus removal) | directly after treatment of the vein (Day 0)
  Society Interventional Radiology (SIR) Grad II Lyse (50-95 % thrombus removal) or greater at the end of the procedure including adjunctive treatments
Vilallta score | Day 0, month 1 and 6
  Score for post thrombotic syndrome (PTS) assessing 5 subjective symptoms (pain, cramps, heaviness, paresthesia, pruritus) and 6 clinical signs (pretibial edema, skin induration, hyperpigmentation, redness, venous ectasia, pain on calf compression) with a 4-point scale from 0 (not present) to 3 (severe).
Venous clinical severity score (VCSS) | Day 0, month 1 and 6
  Score of 10 parameters each assessed by severity 0-3.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Lichtenberg, MD, Principal Investigator — Klinikum Hochsauerland GmbH
Locations (1):
- Klinikum Hochsauerland GmbH, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No
It is not planned to share IPD